CLINICAL TRIAL: NCT04320537
Title: Brain Neurochemical Profile During Marijuana Abstinence
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: Scott E. Lukas, PhD, McLean Hospital (Unknown)
Responsible Party: Principal Investigator, Chun S. Zuo, Assistant Professor, Mclean Hospital
Other Study IDs: 2016P001508
Record Dates: First submitted 2020-03-22; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Brain Metabolic Changes During Marijuana Abstinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MJ user: non-treatment-seeking chronic heavy marijuana (MJ) users of both sexes and all ethnicities between the ages of 21-40 years who are willing to follow the study protocol and abstinence from marijuana for three weeks
  Interventions: Other: abstinence from use of marijuana and other abused drugs
- Control: age- and sex-matched healthy control participants who are willing to follow the study protocol and remain in the study for three weeks
  Interventions: Other: abstinence from use of marijuana and other abused drugs

INTERVENTIONS:
Other: abstinence from use of marijuana and other abused drugs — abstinence from use of marijuana use and other abused drugs

SUMMARY:
We have interviewed more than 120+ candidates and recruited 44 chronic marijuana users and 11 non-user healthy controls: 26 of the 44 MJ users actually participated in the study, 6 of the 26 MJ participants dropped out after their baseline magnetic resonance (MR) visits and the remaining 20 participants completed the study protocol, namely completed three MR visits for measurement of brain metabolites (baseline, day 7, and day 21); among the 11 healthy controls, 10 completed the study protocol. We are currently analyzing collected data and preparing manuscripts for peer reviewed journals.

DETAILED DESCRIPTION:
Marijuana (MJ) is the most widely used illicit drug in the US among young adults. A majority of those who enter treatment for MJ dependence relapse. However, the mechanism of action of MJ on brain neurochemistry, especially in connection with the reported withdrawal symptoms, is still not well understood. We hypothesized that brain gamma aminobutyric acid (GABA) and glutamate (glu) fluctuate during the transition between active exposure, early abstinence (1-2 days since last use), and prolonged abstinence (7 days and more), and an imbalance of GABA and glu during MJ abstinence was the metabolic source of the aforementioned withdrawal symptoms that make MJ abstinence so difficult for many individuals. The investigator's specific aims were to measure MJ abstinence related changes in levels of GABA and glu and to correlate the changes in GABA and glu with MJ withdrawal symptoms and clinical measures at baseline, day 7, and day 21 into abstinence. The MR measures were conducted at 3 tesla and the abstinence was verified by urinary tetrahydrocannabinol (THC) levels.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants must be 21-40 years of age. 2. Women must not be pregnant, planning to get pregnant, or lactating. 3. Individuals must meet criteria of chronic, heavy use of marijuana to be enrolled in the group of MJ-users. Namely, participants in this group may, but do not have to, meet DSM-5 criteria for cannabis use disorder based on the Structured Clinical Interview for DSM Disorders (SCID-5) and they have to have had at least one years of reported use of four out of seven days per week, or greater than 25 episodes per month. An "episode" is defined as an occasion of smoking separated by at least one hour from another "episode." 4. Participants must be able to comply with the study protocol, willing to remain abstinent during the 3-week period, willing to limit amounts of alcohol and tobacco consumption during the study period, and willing to commit the time to participate in the study. 5. Participants must be able to provide written informed consent. 6. Participants must be able and willing to complete questionnaires during various visits.

Exclusion Criteria:

* 1. Individuals with significant and symptomatic medical or neurological co-morbidity, such as chronic fatigue syndrome or fibromyalgia, or any current Axis I Psychiatric Disorder, severe medical conditions such as multiple sclerosis, anemia, cancer, cirrhosis, heart disease, or kidney disease, or history of head trauma resulting in loss of consciousness requiring hospital evaluation. 2. Individuals who have been on atypical antipsychotic medications, sleeping medications, or steroid/testosterone. 3. Individuals must not have been on stimulant medications or antidepressant medications including Selective Serotonin Reuptake Inhibitors (SSRIs), for at least one year. 4. Individuals must not currently hold a medical marijuana certificate. 5. Individuals who, in the Principal Investigator's judgment, will not likely be able to comply with the study protocol. 6. Individuals meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for current substance use disorder other than MJ 7. Individuals who have any lifetime regular use of cocaine, stimulants, or hallucinogens more than twice monthly 8. Individuals who smoke more than 10 tobacco cigarettes daily 9. Individuals who consume more than two alcoholic drinks per day, on average, or report binge drinking (4 or more drinks for women, 5 or more drinks for men).

In addition to the above criteria, the following exclusion criteria apply for subjects participating in this MR study:

MR Exclusion Criteria:

1. Contraindication to MR scanning, including claustrophobia.
2. Individuals unable to comply with instructions or procedures of study.
3. Presence of metal pins or braces in subject.
4. Evidence of structural brain abnormalities on brain MRI. (Inclusion Criteria and Exclusion Criteria for the subjects including controls have been stated in above section D Research Design and Methods)

Ages: 21 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Participants were recruited without regard to sex, race, or ethnicity. Based on prior research studies at McLean Hospital, in the northwest suburbs of Boston, we expect the number of men and women to be approximately equal, and about 5-15% of subjects to be African-American or Hispanic. Overall, these distributions are not very different from the population statistics for the Greater Boston Area of 82.6% White, 8.3% African American, 6.3% Asian, and 2.8% of other ethnic or racial backgrounds based on 2014 census.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Brain Neurochemical Profile during Marijuana Abstinence | three weeks
  brain metabolites correlated with withdrawal symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Chun Zuo, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Will follow NIH policy